CLINICAL TRIAL: NCT05635643
Title: A Phase 1 Study of CHS-114 in Participants With Advanced Solid Tumors
Brief Title: Study of CHS-114 in Participants With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Coherus Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SRF114-101
Record Dates: First submitted 2022-11-14; First posted 2022-12-02 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Advanced Solid Tumor; Head and Neck Squamous Cell Carcinoma
Keywords: metastatic solid tumors; advanced solid tumors; Phase 1; SRF114; CCR8; safety; efficacy; immunotherapy; cancer; immuno-oncology; CHS-114
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Neoplasms | interventions — toripalimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm 1a: CHS-114 Dose Escalation (Experimental): Arm 1 monotherapy dose escalation portion of the study will evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics, and preliminary efficacy of CHS-114 as monotherapy in up to 25 participants with advanced solid tumors, to determine the recommended dose for expansion (RDE).
  Interventions: Drug: CHS-114
- Arm 1b: CHS-114 Dose Expansion (Experimental): Arm 1b monotherapy expansion will evaluate the safety, tolerability, PK, pharmacodynamics, and efficacy of CHS-114 monotherapy at 2 dose levels (potential recommended dose for expansion RDE in up to 5 participants in each dose level with Head and Neck Squamous Cell Carcinoma (HNSCC).
  Interventions: Drug: CHS-114
- Arm 2: CHS-114 + toripalimab Dose Escalation (Experimental): Arm 2 dose escalation will evaluate the safety, tolerability, PK, pharmacodynamics, and efficacy of CHS-114 in combination with toripalimab at 2 RDE levels in up to 6 participants in each dose level with HNSCC.
  Interventions: Drug: CHS-114; Drug: toripalimab
- Arm 3: CHS-114 + toripalimab Dose Expansion (Experimental): Arm 3 dose expansion will evaluate the safety, tolerability, PK, pharmacodynamics, and efficacy of CHS-114 in combination with toripalimab at 2 RDE levels in up to 20 participants in each dose level with HNSCC.
  Interventions: Drug: CHS-114; Drug: toripalimab

INTERVENTIONS:
Drug: CHS-114 — CHS-114
Drug: toripalimab — toripalimab-tpzi
  Other Names: Loqtorzi
  Arms: Arm 2: CHS-114 + toripalimab Dose Escalation; Arm 3: CHS-114 + toripalimab Dose Expansion

SUMMARY:
This is a Phase 1, open-label, first-in-human, dose-escalation and expansion study of CHS-114, a monoclonal antibody that targets CCR8, as a monotherapy in patients with solid tumors.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, first-in-human, dose-escalation and expansion study of CHS-114, a monoclonal antibody that targets CCR8, as a monotherapy in participants with advanced solid tumors, that will be conducted in 3 parts:

* Arm 1a: CHS-114 monotherapy dose-escalation portion of the study will enroll approximately 25 participants with advanced solid tumors.
* Arm 1b: CHS-114 monotherapy expansion cohort(s) will evaluate the safety, efficacy, tolerability, pharmacokinetics, and pharmacodynamics of CHS-114 in indication specific cohort(s). Up to approximately 10 participants will be enrolled.
* Arm 2: CHS-114 + toripalimab combination dose-escalation portion of the study will evaluate the safety, efficacy, tolerability, pharmacokinetics, and pharmacodynamics of CHS-114 in combination with toripalimab in indication specific cohort(s). Up to approximately 6-12 participants will be enrolled.
* Arm 3: CHS-114 + toripalimab combination dose-expansion portion of the study will evaluate the safety, efficacy, tolerability, pharmacokinetics, and pharmacodynamics of CHS-114 in combination with toripalimab in indication specific cohort(s). Up to approximately 40 participants will be randomized to two dosing arms.

ELIGIBILITY:
Key Inclusion Criteria - Arms 1a, 1b, 2, and 3

* Participants must be ≥ 18 years of age.
* For Arm 1a only, locally advanced or metastatic (Stage IV) solid tumor that has progressed during or after standard therapy and for whom no available therapies are appropriate (based on the judgment of the Investigator).
* At least 1 measurable lesion per RECIST 1.1.
* Lesions previously treated with radiation or other forms of locoregional therapy must show radiographic evidence of disease progression to be used as a target lesion.
* For Arms 1a, 1b, and 2 only, washout period from the last dose of previous anticancer therapy (chemotherapy, biologic, or other investigational agent) to the initiation of study drug must be > 5 times the half-life of the agent or > 21 days (whichever is shorter).
* Resolution of non-immune-related AEs secondary to prior anticancer therapy (excluding alopecia and peripheral neuropathy) to ≤ Grade 1 per NCI-CTCAE version 5.0 or higher, and complete resolution of immune-related AEs secondary to prior checkpoint inhibitor therapy.
* Serum creatinine clearance ≥ 30 mL/min per Cockcroft-Gault formula.
* Total bilirubin ≤ 1.5 × ULN (≤ 3 × ULN if elevated because of liver metastases or documented Gilbert's syndrome).
* Aspartate aminotransferase/serum glutamic oxaloacetic transaminase (AST/SGOT) and alanine aminotransferase/serum glutamic pyruvic transaminase (ALT/SGPT) < 2.5 × ULN or < 5 × ULN for patients with known liver metastases.
* Adequate hematologic function, defined as absolute neutrophil count ≥ 1.0 × 10^9/L, hemoglobin ≥ 8.0 g/dL, and platelet count ≥ 75 × 10^9/L.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Ejection fraction ≥ 50%, as measured by echocardiogram, multigated acquisition scan, nuclear stress test, or equivalent modality.
* Willingness of male and female patients who are not surgically sterile or postmenopausal to use medically acceptable methods of birth control for the duration of the study treatment period, including 90 days after the last dose of CHS-114, 4 months after the last dose of toripalimab; male patients must refrain from donating sperm during this period. Sexually active men, and women using oral contraceptive pills, should also use barrier contraception. Azoospermic male patients and women of childbearing potential who are continuously not heterosexually active are exempt from contraceptive requirements.

Additional Inclusion Criteria - Arms 1b and 2 only

* Histologically or cytologically confirmed advanced or metastatic HNSCC that has progressed during or after a platinum-based chemotherapy and/or a programmed cell death receptor (PD)-1 or PD ligand 1 (PD-L1) targeting agent (separately or in combination therapy).
* Metastatic or locoregionally recurrent HNSCC malignancy that is incurable by surgery or radiotherapy.
* Arm 1b only, participants must have tumor tissue that is accessible for pretreatment and on-treatment tumor biopsy in the opinion of the Investigator and be willing and consent to undergo pretreatment and on-treatment biopsies per protocol.

Additional Inclusion Criteria - Arm 3 only

* Histologically or cytologically confirmed locally advanced or metastatic HNSCC (primary tumor location of oral cavity, oropharynx, hypopharynx, or larynx). Participants may not have a primary tumor site of nasopharynx (any histology).
* Participants should have been treated with anti-PD-1/PD-L1-directed systemic therapy for incurable recurrent, advanced, or metastatic disease and experienced progressive disease. targeting agent (separately or in combination therapy).
* Metastatic or locoregionally recurrent HNSCC malignancy that is incurable by surgery or radiotherapy.
* Consent to provide HPV status assessed by p16 and results from baseline PD-L1 IHC assay score.
* Consent to provide tumor tissue samples is required for enrollment.

Key Exclusion Criteria - Arms 1a, 1b, 2, and 3

* Previously received an anti-CCR8 antibody or anti-CCR8 targeted therapy.
* History of Grade 4 allergic or anaphylactic reaction to any monoclonal antibody therapy or any excipient in the study drugs.
* Major surgery within 4 weeks prior to Screening.
* Unstable or severe uncontrolled medical condition (eg, unstable cardiac function, unstable pulmonary condition including pneumonitis and/or interstitial lung disease, uncontrolled diabetes, symptomatic fistula) or any important medical illness or abnormal laboratory finding that would, in the Investigator's judgment, increase the risk to the patient associated with his or her participation in the study.

Additional Exclusion Criteria - Arms 1b and 2 only

* Received > 4 prior systemic regimens for advanced/metastatic disease.
* Nasopharyngeal carcinoma or nasal cavity malignancies other than HNSCC (eg, adenocarcinoma and variants, neuroendocrine tumors, mucosal melanoma).
* Receiving chronic anti-coagulation therapy (eg, warfarin, enoxaparin) that cannot be safely discontinued temporarily for the required biopsies (only for patients who provide tumor biopsies).

Additional Exclusion Criteria - Arm 3

• Received ≥ 2 prior systemic regimens for advanced/metastatic disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
[Arms 1a, 1b, and 2] Rate of Dose Limiting Toxicity (DLT) | Assessed during first 21 days of treatment
  Evaluation of rate of DLT of CHS-114 as a monotherapy, or in combination with toripalimab
[Arm 2] Summary of adverse events (AEs) based on treatment emergent AEs (TEAEs), anti-drug antibodies (ADA), and laboratory values. | Up to 24 months
  Safety and tolerability of CHS-114 in combination with toripalimab,
[Arm 3] Safety and tolerability of CHS-114 in combination with toripalimab will be assessed by summarizing AEs and will be based on TEAEs as assessed by Common Terminology Criteria for Adverse Events (CTCAE) v5.0 or higher. | Up to 24 months
  Safety and tolerability of CHS-114 in combination with toripalimab

SECONDARY OUTCOMES:
[Arms 1a and 1b] Summary of AEs based on TEAEs. | Up to 24 months
  Safety and tolerability of CHS-114 as monotherapy will be assessed by summarizing AEs and will be based on TEAEs as assessed by CTCAE v5.0 or higher.
[Arms 1a and 1b] ADAs to CHS-114 | Up to 24 months
  Serum will be collected and assessed for the development of ADAs to CHS-114
[Arms 1a, 1b, 2, and 3] PK of CHS-114 | Up to 24 months
  Serum concentrations of CHS-114 will be collected and analyzed to evaluate the PK of CHS-114 and in Arms 2 and 3, toripalimab.
[Arms 1a, 1b, 2, and 3] Confirmed objective response rate (ORR) | Up to 24 months
  Confirmed objective response rate (ORR) based on RECIST v1.1
[Arms 1a, 1b, 2, and 3] Duration of response (DoR) | Up to 24 months
  Duration of response (DoR) based on RECIST v1.1. DoR is defined as the time from the first documented response (CR or PR) to documented disease progression as determined by RECIST v1.1 or death.
[Arms 1a, 1b, 2, and 3] Disease control rate (DCR) | Up to 24 months
  DCR based on RECIST v1.1. DCR is defined as the percentage of patients with CR, partial PR, or stable disease lasting a minimum of 12 weeks.
[Arms 1a, 1b, 2, and 3] Progression-free survival (PFS) | Up to 24 months
  PFS based on RECIST v1.1. PFS is defined as the time from the first treatment on study with study drug to documented disease progression as determined by RECIST v1.1 or death.
[Arms 1a, 1b, 2, and 3] Changes in FOXP3 levels in participants undergoing pretreatment and on-treatment tumor biopsies | Up to 24 months
  Cellular FOX3P expression within the tumor will be collected and analyzed in participants who are undergoing pretreatment and on-treatment biopsies

CONTACTS AND LOCATIONS:
Overall Officials: Koho Izuka, MD, Study Director — Coherus BioSciences
Locations (16):
- United States (16):
  - Hoag Memorial Hospital, Newport Beach, California
  - FOMAT Medical Research, Oxnard, California
  - Stanford Cancer Center, Palo Alto, California
  - SCRI Lake Nona DDU (FL Cancer Specialists), Orlando, Florida
  - Emory Winship Cancer Institute, Atlanta, Georgia
  - Hope & Healing Cancer Services, Hinsdale, Illinois
  - University of Louisville, Louisville, Kentucky
  - University of Maryland Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute - Karmanos Cancer Center, Detroit, Michigan
  - Washington University, St Louis, Missouri
  - University of Cincinnati, Cincinnati, Ohio
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - START- San Antonio, San Antonio, Texas
  - START Mountain, West Valley City, Utah
  - University of Washington/Fred Hutchinson Cancer Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang X, Kapoor VN, Chin DJ, Klakamp SL, Baruffaldi F, Mohan JF, Haines R, Dulak A, Panduro M, Ren Y, Masia R, Hill JA, LaVallee TM, Rajasekaran N. CHS-114: an afucosylated anti-CCR8 monoclonal antibody that selectively depletes intratumoral Treg cells and induces antitumor immune responses. Mol Cancer Ther. 2025 Dec 22. doi: 10.1158/1535-7163.MCT-25-0367. Online ahead of print. PMID 41423415